CLINICAL TRIAL: NCT05622630
Title: Prospective Randomized Study of Physical Therapy in Patients With Diabetic Polyneuropathy
Brief Title: Study of Physical Therapy in Patients With Diabetic Polyneuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Paracelsus Harz Clinic Bad Suderode. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ParacelsusHCBS 51/15
Record Dates: First submitted 2020-09-28; First posted 2022-11-18 (Actual); Last update posted 2022-11-18 (Actual); Status verified 2022-09

CONDITIONS: Diabetic Polyneuropathy
MeSH Terms: conditions — Diabetic Neuropathies | interventions — Baths

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Four-cell bathroom (Active Comparator): Four-cell bath:Treatment with direct current
  Interventions: Procedure: Four-cell bath
- Gravel bath (Active Comparator): Gravel bath:In this procedure, the patients are given a footbath with heated stones (granules) of different sizes for a period of 20 minutes, during which the patients are encouraged to move their feet (and, if applicable, hands) evenly.
  Interventions: Procedure: Gravel bath

INTERVENTIONS:
Procedure: Four-cell bath — Four-cell bath:Treatment with direct current
  Arms: Four-cell bathroom
Procedure: Gravel bath — Gravel bath:In this procedure, the patients are given a footbath with heated stones (granules) of different sizes for a period of 20 minutes, during which the patients are encouraged to move their feet (and, if applicable, hands) evenly.
  Arms: Gravel bath

SUMMARY:
Sensorimotor diabetic polyneuropathy is a common and serious complication of longstanding diabetes mellitus. The therapeutic options are limited (pain therapy, antidepressants, physical measures using direct current such as two- / four-cell baths). In the present study, for the first time, after positive data from a pilot study, it is to be checked whether the effectiveness of an existing therapy can be extended by treatment with heated granulate stones in the rehabilitation setting.

DETAILED DESCRIPTION:
The central aspect of this study is the proof of the effectiveness of the therapeutic treatment of diabetic polyneuropathy with heated granulate stones.

Subsequent information from the study doctor and the patient's written consent will remove the sociodemographic relationships from the standards of the Paracelsus Harz Clinic Bad Suderode. Behavioral behavior and sporting behavior among those affected, as well as the course of the disease, are treated using a questionnaire. Furthermore, medical parameters (echocardiographic parameters, penalties, weight, BMI, waist-hip ratio, blood glucose, HbA1c, total cholesterol, HDL cholesterol, LDL cholesterol, triglyceride, etc.) are determined.

A randomization list was created for randomization, with the randomization algorithm assigning patient IDs to the two treatment groups. Randomization takes place using previously sealed, opaque and consecutively numbered envelopes.

After randomization at time T0 (before the first treatment) and T1 (after the last treatment), the patients receive a questionnaire (see appendix) in which they should state the symptoms, how long they have existed and the assessment of the intensity. The assessment of the intensity is based on a spectrum from 1 = minor complaints to 6 = severe complaints.

Quality of life is measured using the SF-12 questionnaire, and anxiety and depression using the HADS questionnaire are also measured at time points T0 and T1.

Long-term ECGs are performed to determine the heart rate variability at the beginning and at the end of the rehabilitation measure.

A vibration sensation test with the tuning fork (8/8 scale) according to Rydel-Seiffer on the metatarsophalangeal joint of the big toe, the inner ankle and the tibial tuberosity is also carried out at time T0 and T1.

In the study group, the patients receive a foot bath treatment with heated stones of different sizes three times a week for a period of 20 minutes. In the control group, therapy with direct current (four-cell bath) is carried out. The study population consists of patients from the Paracelsus Harz Clinic Bad Suderode who are undergoing rehabilitation due to cardiovascular diseases and / or diabetes mellitus.

It is planned to start at time T0 with n = 34 rehabilitation patients in the basement and in the KG. Even with a pessimistically estimated drop-out rate of 20% in the course of the study at time T1 (after completion of the rehabilitation measure), n = 28 test persons per group should still be available. This means that there are enough cases for stratifying analyzes. With this case number planning, the criteria of a case number planning carried out are met. Based on a planned power of the investigation of 80% (α = 0.05) with a drop-out of 20%, this calculation resulted in a sample size of at least n = 28 subjects per group.

ELIGIBILITY:
Inclusion Criteria:

* Age> 18 years of age
* diabetic polyneuropathy
* Inpatient stay in the Paracelsus Harz Clinic Bad Suderode

Exclusion Criteria:

* Lack of consent
* Infections on the extremities to be bathed
* Skin damage on the extremities to be bathed
* Pacemaker or ICD implantation
* Metal (e.g. osteosynthesis materials) in the parts of the body to be bathed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2019-08-13 (Actual); Primary Completion 2021-08-24 (Actual); Study Completion 2022-03-16 (Actual)

PRIMARY OUTCOMES:
Vibration sensation test | baseline
  Vibration sensation test with the tuning fork (8/8 scale) according to Rydel-Seiffer on the wrist, metatarsophalangeal joint of the big toe, inner ankle and the tibial tuberosity
Vibration sensation test | day 20
  Vibration sensation test with the tuning fork (8/8 scale) according to Rydel-Seiffer on the wrist, metatarsophalangeal joint of the big toe, inner ankle and the tibial

CONTACTS AND LOCATIONS:
Locations (1):
- Paracelsus-Harz-Clinic Bad Suderode, Quedlinburg, Saxony, Germany

REFERENCES:
- [Derived] Strobel A, Laputsina V, Heinze V, Schulz S, Wienke A, Reer M, Schlitt A. Nonpharmaceutical treatment of distal sensorimotor polyneuropathy in diabetic patients: an unblinded randomized clinical trial. BMC Complement Med Ther. 2025 Mar 6;25(1):93. doi: 10.1186/s12906-025-04830-0. PMID 40050870